CLINICAL TRIAL: NCT00375115
Title: Efficacy of Sambucol on the Length of Time to Resolution of Influenza Illness
Brief Title: Efficacy of Sambucol in the Treatment of Influenza
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Razei Bar industries Ltd. (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 360HMO-CTIL
Record Dates: First submitted 2006-09-10; First posted 2006-09-12 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2007-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — black elderberry extract

INTERVENTIONS:
Drug: Sambucol

SUMMARY:
The trial will examine the efficacy of sambucol in the treatment of influenza. The primary efficacy endpoint will be the length of time to resolution of influenza illness.The double blind trial will be conducted at the Personnel Clinic, and at the Clinical virology Unit, Hadassah University Hospital, and will include 100 patients with laboratory-confirmed influenza infection, 50 in the sambucol and 50 in the placebo study arm.

DETAILED DESCRIPTION:
The trial will be conducted at the Personnel Clinic, and at the Clinical virology Unit, Hadassah University Hospital.

Candidates for participation in the trial :

Patients who will present at the clinic with influenza-like symptoms; men and women ages 20 yrs- 65 yrs who will sign written informed consent

Excluded from the trial will be:

* Pregnant women or women who cannot exclude pregnancy.
* Patients with diabetes.
* Immune-suppressed patients, including patients taking immunosuppressive drugs.
* Patients with renal failure.
* Patients who received the recent influenza vaccine.

The study participants will receive treatment (either Sambucol or placebo) for five days. The follow-up period will be 10 days. All patients initially included in the trial will be followed for 10 days.

Inclusion criteria:

* Fever ≥ 380C.
* The presence of at least one of the following respiratory symptoms: cough, sore throat, nasal congestion/ runny nose.
* The presence of at least one of the following systemic symptoms: headache, fatigue, myalgia, chills/sweats, malaise.

Study Patients A total of 100 patients with laboratory-confirmed influenza infection will be included in the study (50 in each study arm).

This calculation is based on the expected percentage of recovery within 3 days from initial treatment (allowing that 80% of patients given the active component will show improvement as opposed to 50% of placebo patients).

Assuming that 50% of the patients presenting with influenza-like illness will have a laboratory-confirmed influenza infection, a total number of 200 patients is expected.

The primary efficacy endpoint will be the length of time to resolution of influenza illness (defined as the period from start of study drug to the relief of symptoms).

Study design:

1. Patients presenting at the clinic with the above indicated inclusion criteria will be referred by the clinic nurse to a physician to establish the diagnosis
2. The temperature, the presence and severity of influenza symptoms including cough, nasal obstruction, sore throat, fatigue, headache, myalgia will be recorded on a four-point scale (0-absent, 1-mild, 2-moderate, 3-severe). Patients will also record their ability to do their normal activities, overall health status, and sleep quality on a ten-point scale (0-unable or worst, to 10-fully able, best)
3. For influenza detection, nose and throat swabs will be collected at baseline.
4. Patients will be randomly assigned to receive either Sambucol or placebo (15 cc 4 times daily for 5 days).
5. Patients will be instructed that relief medications (Acamol /Optalgin) will be taken only as required, and that their use should be recorded.
6. The follow-up will include all the parameters (see "2") recorded daily at days 1-5, at day 7, and at day 10.
7. Compliance with the study drug will be recorded.
8. In case the patient's condition deteriorates, the patient will be examined at the clinic to rule out the presence of complications (such as pneumonia, sinusitis, or bronchitis).
9. Statistical analysis will include the duration and severity of the symptoms as well as the use of relief medications.

Laboratory diagnosis of influenza infection:

Combined nose and throat specimens will be tested for the presence of influenza virus at the Clinical Virology Unit by real-time PCR, following viral RNA extraction, using the TaqMan ABI 7900 instrument. Primers and fluorescent probes specific for influenza A and B viruses will be employed in a multiplex reaction.

Specimens found positive for influenza by real-time PCR will be further subjected to influenza culture on MDCK cells.

The recovered influenza viruses will be subtyped by hemagglutination inhibition, using specific antisera obtained from the WHO, or by multiplex reverse transcription (RT)- PCR reaction, using specific primers for influenza B as well as for the different influenza A H and N.

ELIGIBILITY:
Inclusion Criteria:

* Fever ≥ 380C.
* The presence of at least one of the following respiratory symptoms: cough, sore throat, nasal congestion/ runny nose.
* The presence of at least one of the following systemic symptoms: headache, fatigue, myalgia, chills/sweats, malaise.

Exclusion Criteria:

* Pregnant women or women who cannot exclude pregnancy.

  * Patients with diabetes.
  * Immune-suppressed patients, including patients taking immunosuppressive drugs.
  * Patients with renal failure.
  * Patients who received the recent influenza vaccine.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-09; Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The length of time to resolution of influenza illness

CONTACTS AND LOCATIONS:
Overall Officials: Dana G Wolf, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel